CLINICAL TRIAL: NCT05033808
Title: Epirubicin for the Treatment of Sepsis & Septic Shock
Acronym: EPOS-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jena University Hospital (Other)
Collaborators: Ruhr University of Bochum (Other); University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPOS_ZKSJ0134; 2021-002300-12 (EudraCT Number); 01EN2001 (Other Grant/Funding Number: German Federal Ministry of Education and Research); DRKS00025884 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2021-08-04; First posted 2021-09-05 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Sepsis
Keywords: epirubicin; disease tolerance; myelotoxicity; pilot study
MeSH Terms: conditions — Sepsis | interventions — Epirubicin

STUDY DESIGN:
Intervention Model Description: Sequential dose escalation with three dosing groups and placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study medication is provided in colored infusion bags with additional covers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Administration of NaCl i.v. as placebo once.
  Interventions: Drug: Placebo
- Epirubicin Phase I (Experimental): Administration of epirubicin i.v. 3.75 mg/m2 once.
  Interventions: Drug: Epirubicin
- Epirubicin Phase II (Experimental): Administration of epirubicin i.v. 7.5 mg/m2 once.
  Interventions: Drug: Epirubicin
- Epirubicin Phase III (Experimental): Administration of epirubicin i.v. 15 mg/m2 once.
  Interventions: Drug: Epirubicin

INTERVENTIONS:
Drug: Epirubicin — Epirubicin is given once over 15 Minutes via a central line
  Arms: Epirubicin Phase I; Epirubicin Phase II; Epirubicin Phase III
Drug: Placebo — NaCl is given once over 15 Minutes via a central line
  Arms: Placebo

SUMMARY:
The study will assess the safety of low doses of epirubicin in sepsis patients. Therefore the study will look for side effects in patients treated with low dose epirubicin compared to control patients.

In animals, low dose epirubicin has been shown to induce tolerance to infection and increase survival in septic mice.

The study will also look for positive effects on organ function in humans. The investigators hypothesize that low-dose epirubicin can be used therapeutically to improve the disease course and lessen mortality of patients with sepsis. In a first step, the investigators aim at proving that low-dose epirubicin can safely be administered to sepsis patients and will perform a dose-escalation multi-center trial.

DETAILED DESCRIPTION:
There are two ways for organism to deal with infection. Resistance, which means elimination of infectious microorganisms by the immune system, is widely recognized. It can be supported by antibiotic medication and surgical or interventional drainage of an infectious focus. The other response is tolerance, which means limiting organ damage without fighting the infection itself. Its importance has become more clearly recently, but so far there are no therapeutic interventions to support this mechanism.

Epirubicin is a chemotherapeutic substance used to treat cancer. In animal experiments, it has been shown that doses much lower than the ones used in oncology, can induce tolerance in infected animals. Animals treated with epirubicin survive an infectious dose that kills animals not treated with epirubicin. Before this approach can be studied in a large group of sepsis patients, it is necessary that epirubicin in low doses can be safely used in this population.

Therefore in this study, septic patients will be treated with low doses of epirubicin and systematically assessed for serious side effects. Some patients will be treated with placebo for comparison. The trial will be conducted as a dose escalation study with three groups. This means that the first group of patients will receive only a quarter of the dose shown to be effective in animal experiments. Only if no serious side effects are observed will the dose be increased in the second group and again in the third group.

In addition, the study will look for signs of beneficial effects on organ function in human patients with sepsis, pharmacokinetics of epirubicin in sepsis patients and changes in the inflammatory response.

The investigators hypothesize that low-dose epirubicin can be used therapeutically to improve the disease course and lessen mortality of patients with sepsis. In a first step, the investigators aim at proving that low-dose epirubicin can safely be administered to sepsis patients and will perform a phase IIa dose-escalation multi-center trial.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the ICU with sepsis or septic shock, diagnosed within the previous 24 hours

Exclusion Criteria:

* Leukopenia/Neutropenia/Thrombocytopenia-prior or upon inclusion (Leucocyte Count <4000/μL; Neutrophile/ platelets Count below Lower Limit of Normal).
* Weight >135 kg/BMI >45.
* Active neoplasia.
* History of chemotherapy.
* Hypersensitivity to epirubicin
* History of bone marrow or solid organ transplantation.
* Immunosuppressive therapy.
* Acute severe infection within 4 weeks prior to admission (Hospitalization or admission to higher level clinical care facility for infection).
* Chronic infection.
* Cardiomyopathy with a documented ejection fraction <30% or AICD (automatic internal cardioverter defibrillator) implantation.
* Acute liver failure following the European Association for the Study of the Liver definition as International Normalized Ratio (INR) >1.5 and elevation of transaminases > 3 times of the upper normal limit (2).
* Pregnancy during all trimesters/breast-feeding.
* Chronic mechanical ventilation dependency.
* Cystic fibrosis.
* Concomitant medication with Verapamil or Cimetidine.
* Prior enrollment in this study.
* Participation in another clinical intervention trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with myelotoxicity | Up to 14 days after administration of study drug
  Neutropenia or thrombocytopenia of grade 3 or 4 (neutrophiles <1,000μL or platelets <50,000/μL) at two consecutive study visits up to day 14 accompanied by neutropenia or thrombocytopenia of grade 2, 3 or 4 (neutrophiles <1,500μL or platelets <75,000/μL) at both study visits and accompanied by an IPF (immature platelet fraction) below 2.5% at one or two of the consecutive study visits.

SECONDARY OUTCOMES:
Survival at day 14, 28 and 90 | 14, 28 and 90 days
  Survival
SOFA score | Up to 14 days after administration of study drug
  SOFA (sequential organ failure assessment) on days of assessment, mean total SOFA and SOFA changes over time
Cardiotoxicity | 7 days after administration of study drug
  Ejection fraction measured via TTE (trans-thoracic echocardiography)
"Success" rate | 3 days after administration of study drug
  Decrease of procalcitonin (PCT) serum concentration by 80% or more of its intra-individual peak value or to 0.5 μg/L or lower within 72 hours after randomization
Adverse events | Up to 90 days after administration of study drug
  Overall rate of adverse and severe adverse events. The the frequency of other typical side effects (diarrhea, mucositis, alopecia, nausea and vomiting).
Quality of life assesed by the SF-36 questionaire | At follow up 90 days after administration of study drug
  The short Form 36 Health Questionnaire (SF-36) contains 36 questions on quality of life. From the answers a Physical Component Summary (PCS) and a Mental Component Summary (MCS) are calculated, both ranging approximately from 0 (severe disability) up to 80 (absence of disability).
Fluid balance and urine output | Up to 14 days after administration of study drug
  Assessment of fluid balance and urine output
Need for renal replacement therapy | Up to 14 days after administration of study drug
  Use of renal replacement therapy for chronic or acute kidney failure
Oxygenation index (paO2/FiO2) | Up to 14 days after administration of study drug
  The ratio of arterial oxygen partial pressure and the fraction of inhaled oxygen will be calculated. For patients receiving conventional low flow oxygen FiO2 will be estimated based on a predefined table.
Need for respiratory support | Up to 14 days after administration of study drug
  The highest level of respiratory support will be documented.
Need for catecholamines and inotropes | Up to 14 days after administration of study drug
  For all catecholamines and inotropes the highest daily rate administerd for at least one hour will be documented.

OTHER OUTCOMES:
Epirubicin plasma concentrations | At 15minutes and at 1, 2, 3, 6, 12, and 24 hours after administration of study drug
  Epirubicin concentrations in the plasma will be measured using mass-spectrometry
DNA damage | Up to 7 days after administration of study drug
  DNA damage in peripheral mononuclear blood cells (PBMC) will be assessed. Further assessment of molecular parameters from the PBMCs reflecting epirubicin effects on the DNA or damage control pathways will be performed subsequently
Cytokines | Up to 14 days after administration of study drug
  Plasma cytokines will be determined in all patients using Luminex xMAP or alike multiplex technology
Organ damage markers | Up to 14 days after administration of study drug
  Non-conventional sensitive organ damage markers (e.g. NGAL) will be measured
Anti-PF4 anti-bodies | Up to 14 days after administration of study drug
  Determination of anti-PF4 (platelet factor 4) anti-bodies
Mitochondrial function | Up to 7 days after administration of study drug
  Molecular parameters for mitochondrial function will be assessed from isolated PBMCs

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Weis, M.D., Principal Investigator — Jena University Hospital
Locations (5):
- Germany (5):
  - Jena University Hospital, Jena, Thuringia
  - University Hospital Knappschafstkrankenhaus Bochum, Bochum
  - University Medicine Greifswald, Greifswald
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Figueiredo N, Chora A, Raquel H, Pejanovic N, Pereira P, Hartleben B, Neves-Costa A, Moita C, Pedroso D, Pinto A, Marques S, Faridi H, Costa P, Gozzelino R, Zhao JL, Soares MP, Gama-Carvalho M, Martinez J, Zhang Q, Doring G, Grompe M, Simas JP, Huber TB, Baltimore D, Gupta V, Green DR, Ferreira JA, Moita LF. Anthracyclines induce DNA damage response-mediated protection against severe sepsis. Immunity. 2013 Nov 14;39(5):874-84. doi: 10.1016/j.immuni.2013.08.039. Epub 2013 Oct 31. PMID 24184056
- [Derived] Thomas-Ruddel D, Bauer M, Moita LF, Helbig C, Schlattmann P, Ehler J, Rahmel T, Meybohm P, Grundling M, Schenk H, Kocher T, Brunkhorst FM, Graler M, Heger AJ, Weis S; EPOS-1 study group; SepNetCriticalCare TrialsGroup. Epirubicin for the Treatment of Sepsis and Septic Shock (EPOS-1): study protocol for a randomised, placebo-controlled phase IIa dose-escalation trial. BMJ Open. 2024 Apr 22;14(4):e075158. doi: 10.1136/bmjopen-2023-075158. PMID 38653508